CLINICAL TRIAL: NCT02097108
Title: One Arm, Open Label, Interventional, Non-comparative Study to Assess Changes in Lipids and Lipoproteins in HIV Infected Women With Hyperlipidemia After Switch From Boosted Protease Inhibitor to Raltegravir
Brief Title: Changes in Lipids and Lipoproteins in HIV Infected Women After Switch From Protease Inhibitor to Raltegravir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_HIV1
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infections
Keywords: HIV infection; Raltegravir; Switch; Hyperlipidemia; Women
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (Other): Patients will be offered to switch their protease inhibitor containing regimen to a raltegravir (400mg twice daily, orally) based regimen while maintaining the same background therapy.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir

SUMMARY:
This is a 24-week, one arm, open-label, interventional, non-comparative multicenter study to evaluate lipid changes in HIV infected women with hyperlipidemia on boosted PI based regimen after switching their boosted PI to raltegravir at standard dosage with 400mg twice daily.

This study aims to study the effect on metabolic profiles by switching hyperlipidemic HIV infected women from a PI based regimen to raltegravir.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection in female patients, age ≥18 years
* Patients receiving antiretroviral therapy consisting of at least 2 antiretroviral agents other than protease inhibitor plus a ritonavir-boosted protease inhibitor (PI) for at least the previous 6 months
* Plasma HIV viral load <50 copies/ml on current boosted PI containing regimen for ≥ 6 months prior to study entry
* Fasting LDL cholesterol >130 mg/dl
* Fasting triglycerides <450 mg/dl

Exclusion Criteria:

* History of virological failure during previous antiretroviral therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — PMU Salzburg
Locations (3):
- Austria (3):
  - PMU Salzburg, Salzburg
  - AKH Wien, Vienna
  - Ottto Wagner Spital, Vienna

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were enrolled at 3 sites in Austria. First patient in was 15.05.2014; last patient in was 23.06.2015.
Groups:
- Raltegravir: Patients will be offered to switch their protease inhibitor containing regimen to a raltegravir (400mg twice daily, orally) based regimen while maintaining the same background therapy.
  Raltegravir
Period: Overall Study
Arm/Group | Raltegravir
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — patient was abroad for 6 months | 1

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients With Low-density Lipoprotein (LDL) Cholesterol Reduction
Description: A reduction of > 5% in the plasma concentration of direct LDL cholesterol from baseline to week 12 or > 10% reduction of total cholesterol or reduction of lipid lowering agents is expected. Reduction of lipid lowering agents is defined as reduction due to amelioration of lipid profiles and does not include reduction due to side effects or other toxicity issues.
Time Frame: baseline to week 12
Population: all patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 11
percentage of participants | 90.9 [58.7 to 99.8]

2. Secondary Outcome: Total Cholesterol Baseline and After 24 Weeks
Time Frame: baseline to week 24
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Raltegravir
Number analyzed (Participants) | 11
mg/dl
  Baseline | 247.55 (21.07)
  24 weeks | 215.7 (28.55)

3. Secondary Outcome: Triglycerides Baseline and After 24 Weeks
Time Frame: baseline to week 24
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Raltegravir
Number analyzed (Participants) | 11
mg/dl
  Baseline | 168.45 (57.08)
  24 weeks | 83.3 (28.94)

4. Secondary Outcome: High-density Lipoprotein (HDL) Cholesterol Baseline and After 24 Weeks
Time Frame: baseline to week 24
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Raltegravir
Number analyzed (Participants) | 11
mg/dl
  Baseline | 58 (14.09)
  24 weeks | 64 (12.75)

ADVERSE EVENTS:
Time Frame: 19 months
Description: All (serious) adverse events occuring during study treatment were collected until 28 days after the end of study treatment.
Arm/Group | Raltegravir
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other